CLINICAL TRIAL: NCT03831074
Title: Posterior Capsule Opacification and Optical Quality of Different Hydrophobic Acrylic Intraocular Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Katharina Kriechbaum, Assoc. Prof. Dr., Medical University of Vienna
Other Study IDs: 933/2011
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Posterior Capsule Opacification

INTERVENTIONS:
Device: Implantation of an intraocular lenses: iMics 1 NY-60 & NY-60G

SUMMARY:
The most frequent long-term complication of cataract surgery remains to be posterior capsule opacification (PCO). During the past decades many new intraocular lenses (IOL) with optimized lens material and design were introduced. We propose a study comparing three acrylic single-piece IOLs with different design and hydrophobic material. All IOLs (Hoya NY-60, HOYA Surgical Optics GmbH; EyeCee One, Nidek Co., Aichi, Japan) are commercially available and are used for routine cataract surgery. In this study a comparison of PCO score of all two IOLs, a comparison of optic quality with wavefront analyses, visual acuity, contrast sensitivity, IOL decentration and tilt, slitlamp examination, fibrosis, glistening intensity (subjectively scored), YAG capsulotomy rate, and safety parameters (IOL related adverse reactions) of the investigated IOLs will be performed. Since PCO develops slowly within years, a long-term follow-up of three years will be necessary.

As those IOLs are currently often implanted IOLs, their performance on PCO development and their optical quality is of high interest for the ophthalmologic community.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract for which phacoemulsification extraction and posterior IOL implantation has planned
* Age 40 and older
* Visual potential in both eyes of 20/30 or better as determined by investigators estimation
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Preceding ocular surgery or trauma
* Relevant other ophthalmic diseases (such as pseudoexfoliation, retinal degenerations, etc.)
* Uncontrolled systemic or ocular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-01-27 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
Posterior capsule opacification | 3 years
  Posterior capsule opacification in the 2 IOLs will be assessed with semi automated quantification of cataract software

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Kriechbaum, Principal Investigator — Medical University of Vienna